CLINICAL TRIAL: NCT02266420
Title: Comparison of Biological Features Between pN0 Triple Negative Breast Tumours With Size < or = 10 mm (pT1a/b) Versus pT1c T2 < or = 30 mm.
Acronym: COCABIO000
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14 SEIN 09
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-08

CONDITIONS: Triple Negative Breast Cancers Without Lymph-node Involvement and < or = 30 mm
Keywords: Triple negative breast cancer; immuno-histochemistery; genomic profiles
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNBC pT1a/b with size < or = 10 mm (Other): Patients with pN0 triple negative breast tumor with size < or = 10 mm (pT1a/b) Study intervention = blood samples collected at initial visit
  Interventions: Procedure: Blood samples of 10 mL
- TNBC pT1c T2 with size <or = 30 mm (Other): Patients with pN0 triple negative breast tumor with size < or = 30 mm (pT1c T2) Study intervention = blood samples collected at initial visit
  Interventions: Procedure: Blood samples of 10 mL

INTERVENTIONS:
Procedure: Blood samples of 10 mL — Blood samples of 10 mL will be collected at initial visit; serum samples will then be stored at the end of the study (-80°C) and may be used for the purpose of further scientific research.

SUMMARY:
This is a prospective, non-randomized and multicenter study designed to compare biological features between pN0 triple negative breast cancer (TNBC) with size ≤ 10 mm (pT1a/b) versus pT1c T2 ≤ 30 mm.

All consecutive patients will be recruited by each investigator after completion of surgery. No modification of standard management according to each investigator center will be done. All patients will then be followed each year during 5 years in order to collect the following events: local and loco regional recurrence, metastatasis, second cancer, death or not and the cause.

At initial visit, a 10 mL blood sample will be collected (= study intervention) and immediately processed for serum storage; all serum samples will be stored at -80°C and may be used for the purpose of further scientific research.

A representative formalin-fixed paraffin-embedded tumor block of all 200 samples will be addressed at the Institut Claudius Regaud for central collection which will consist of one haematoxylin-eosin stained slide for central histological review, up to 15 unstained slides for DNA extraction (after microdissection), and construction of a tissue micro-array (TMA).

Extracted DNA from 100 samples (50 in each group) will then be transferred to Institut Paoli Calmettes, Marseille; extracted DNA will be subjected to array-CGH analysis in order to detect gene copy number alterations such as gains/amplifications/deletions, and to next generation sequencing (NGS; MiSeq, Illumina) using a panel of ~400 genes for mutation detection.

ELIGIBILITY:
Inclusion Criteria:

1. Woman with age ≥ 18 years.
2. Patient who completed surgery for his breast cancer and for which definitive histo-pathological analysis of surgical specimen is available.
3. Invasive breast carcinoma pN0 or pN(i+) with histological tumor size ≤ 10 mm (pT1a/b subgroup) or invasive breast carcinoma with histological tumor size > 10 mm and ≤ 30 mm (pT1c T2 ≤ 30 mm control group).
4. Patient with HER2-negative breast carcinoma: immuno-histochemistry (IHC) score = 0, 1+ or 2+ and in situ hybridization (FISH, CISH, or SISH) negative (local laboratory testing).
5. Patient with ER and PR negative invasive carcinoma (< 1% stained cells by immuno-histochemistry assay) (local laboratory testing).
6. In case of multifocality, the histological size of the largest tumor must be ≤ 10 mm or ≤ 30 mm according to the inclusion subgroup. All lesions must be ER, PR and HER2-negative.
7. In case of breast conserving surgery, clear margins are required.
8. Patient affiliated to a Social Health Insurance in France.
9. Patient information and written informed consent form signed prior to any study specific procedures.

Exclusion Criteria:

1. Patients with any previous malignancy of the breast or other site, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer totally resected.
2. Non-invasive breast carcinoma (i.e. ductal carcinoma in situ exclusively).
3. Inoperable breast invasive carcinoma.
4. Synchronous bilateral breast cancer.
5. Patients who received neo-adjuvant treatment (radiotherapy or chemotherapy or other before surgery).
6. Pregnant or breast-feeding women.
7. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
8. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Biomarker signature for pT1a/b pN0 triple-negative breast cancers versus pN0 triple-negative breast cancers with size > or = 11 mm and < or = 30 mm. | 3 years.
  biomarker signature will be defined from the protein expression of one or several biomarker(s).

SECONDARY OUTCOMES:
Disease free survival. | 7 years.
  Disease Free Survival is defined as the time from inclusion until any recurrence (local or regional), contro-lateral breast cancer, second primary breast cancer, distant metastasis, or death from any cause.
Metastasis Free Survival. | 7 years.
  Metastasis Free Survival is defined as the time from inclusion until distant metastasis or last follow-up news (censored data). All other events are ignored for this endpoint.
Overall survival. | 7 years.
  Overall survival is defined as the time from inclusion until death from any cause or last follow-up news (censured data).
Description and comparison of gene copy number (array-CGH) and gene mutation (targeted NGS) between pT1a/b pN0 triple-negative breast cancer versus pN0 triple-negative breast cancer with size ≥ 11 mm and ≤ 30 mm. | 7 years.

CONTACTS AND LOCATIONS:
Overall Officials: Florence DALENC, Md., Study Chair — Institut Claudius Regaud
Locations (11):
- France (11):
  - Institut de Cancerologie de L'Ouest - Site Paul Papin, Angers
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CH Emile ROUX, Le Puy-en-Velay
  - CHU de LIMOGES - HOPITAL DUPUYTREN, Limoges
  - Institut Paoli Calmettes, Marseille
  - Institut Regional Du Cancer Montpellier, Montpellier
  - Clinique La Croix Du Sud, Quint-Fonsegrives
  - Institut de Cancerologie de L'Ouest - Site Rene Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif